CLINICAL TRIAL: NCT00203541
Title: Effects of a New Antimicrobial Dressing on Wound Healing and Incidence of Sternal Wound Infections in Subjects Who Have Undergone Cardiac Surgical Procedures Requiring Median Sternotomy
Brief Title: Effects of a New Antimicrobial Dressing on Wound Healing and Incidence of Sternal Wound Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Reallocation of funding.
Sponsor: Tyco Healthcare Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 301.18
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-11-19 (Estimated); Status verified 2007-11

CONDITIONS: Surgical Wound Infection
MeSH Terms: conditions — Surgical Wound Infection

INTERVENTIONS:
Device: TELFA™ A.M.D. Island dressing

SUMMARY:
The primary objective of this pivotal study is to determine if a new antimicrobial dressing, applied to the sternal incisions of cardiac surgical subjects, will demonstrate a decreased cumulative incidence rate(CI) of localized, superficial infections at the sternal incisional site as compared to the control group, regular, non-antimicrobial dressing.

ELIGIBILITY:
Inclusion Criteria:

* Sign an informed consent form that has been approved by the Institutional Review Board.
* Adults at least 18 years of age.
* Be undergoing cardiopulmonary bypass surgery with a median sternotomy.
* Be able to return to the study site, if needed, to have the sternal surgical incision site inspected.

Exclusion Criteria:

* Be participating concurrently in another clinical trial that involves an investigational drug or device that would interfere with this study.
* Be in need of a left ventricular assist device.
* Have an active pre-operative infectious process.
* Subject is to receive another topical antimicrobial agent (i.e., Dermabond® Topical Skin Adhesive) other than the study dressing (as assigned by the randomization schedule).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2004-02; Study Completion 2006-06

PRIMARY OUTCOMES:
Decreased cumulative incidence rate of superficial surgical site infections localized at the sternal incision in the treatment group as compared to the control group.

SECONDARY OUTCOMES:
Reduction of microbial log counts at the incisional site in the treatment group compared to the control group; Decreased cumulative incidence of mediastinitis in the treatment group as compared to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Katie Kavounis, MPH, Study Director — Tyco Healthcare/Kendall
Locations (1):
- Duke University, Durham, North Carolina, United States